CLINICAL TRIAL: NCT03654651
Title: The Role of the Microbiome in Blood Glucose Regulation in Response to Peanut Consumption
Brief Title: Peanuts and Glycemic Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: The Peanut Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: use PKE_PEANUT
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Type2 Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evening Peanut Consumption (Experimental): Participants will consume one ounce per day (28 g) of peanuts as an evening snack (i.e., after dinner and before sleep).
  Interventions: Drug: Peanut
- Evening Snack (Active Comparator): Participants will consume an isocaloric higher carbohydrate snack as an evening snack (i.e., after dinner and before sleep).
  Interventions: Drug: High carbohydrate snack

INTERVENTIONS:
Drug: Peanut — Roasted, unsalted peanuts will be purchased from a local grocery store and provided to subjects to consume.
  Arms: Evening Peanut Consumption
Drug: High carbohydrate snack — Whole wheat crackers will be purchased from a local grocery store and provided to subjects to consume with a spread (e.g. cream cheese or margarine).
  Arms: Evening Snack

SUMMARY:
A two-period randomized crossover study will be conducted to determine the effect of peanuts on glycemic control, and elucidate the role of the microbiome in glucose regulation, in individuals with impaired fasting glucose.

DETAILED DESCRIPTION:
A two-period randomized crossover trial will be conducted. Participants will be randomized to receive each treatment for 6 weeks followed by a minimum 4-week wash-out period. During the peanut treatment, participants will consume one ounce per day (28 g) of peanuts as an evening snack. The control treatments will be an isocaloric higher carbohydrate snack consumed after the evening meal. Markers of glycemic control, cardiovascular risk factors and gut health will be assessed at the beginning and the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Impaired fasting glucose at screening (≥ 100 mg/dL).
* BMI ≥20 and ≤40 kg/m2.

Exclusion Criteria:

* Diagnosed diabetes or fasting glucose >126 mg/dl
* Systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
* Prescribed anti-hypertensive, lipid lowering or glucose lowering drugs
* Established cardiovascular disease, stroke, diabetes, liver, kidney or autoimmune disease or inflammatory conditions
* Use of supplements (psyllium, fish oil, soy lecithin, phytoestrogens) and botanicals and not willing to cease for the duration of the study
* Pregnancy or lactation
* Weight loss of >=10% of body weight within the 6 months prior to enrolling in the study
* Smoking or use of any tobacco products
* Allergy to test foods
* Consumption of >14 alcoholic drinks/week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University; Kristina S Petersen, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapp PA, Kris-Etherton PM, Petersen KS. Peanuts or an Isocaloric Lower Fat, Higher Carbohydrate Nighttime Snack Have Similar Effects on Fasting Glucose in Adults with Elevated Fasting Glucose Concentrations: a 6-Week Randomized Crossover Trial. J Nutr. 2022 Jan 11;152(1):153-162. doi: 10.1093/jn/nxab347. PMID 34562081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 267 participants were screened for eligibility
Pre-assignment Details: 51 participants were randomized. One participant withdrew from study before receiving either intervention
Groups:
- Evening Peanut Consumption - Evening Snack Sequence: First intervention:
  Participants will consume one ounce per day (28 g) of peanuts as an evening snack (i.e., after dinner and before sleep).
  Peanut: Roasted, unsalted peanuts will be purchased from a local grocery store and provided to subjects to consume.
  Second intervention:
  Participants will consume an isocaloric higher carbohydrate snack as an evening snack (i.e., after dinner and before sleep).
  High carbohydrate snack: Whole wheat crackers will be purchased from a local grocery store and provided to subjects to consume with a spread (e.g. cream cheese or margarine).
- Evening Snack-Evening Peanut Consumption Sequence: First intervention:
  Participants will consume an isocaloric higher carbohydrate snack as an evening snack (i.e., after dinner and before sleep).
  High carbohydrate snack: Whole wheat crackers will be purchased from a local grocery store and provided to subjects to consume with a spread (e.g. cream cheese or margarine).
  Second intervention:
  Participants will consume one ounce per day (28 g) of peanuts as an evening snack (i.e., after dinner and before sleep).
  Peanut: Roasted, unsalted peanuts will be purchased from a local grocery store and provided to subjects to consume.
Period: First Intervention (6 Weeks)
Arm/Group | Evening Peanut Consumption - Evening Snack Sequence | Evening Snack-Evening Peanut Consumption Sequence
Started | 26 | 25
Completed | 25 | 25
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout Period (2-weeks)
Arm/Group | Evening Peanut Consumption - Evening Snack Sequence | Evening Snack-Evening Peanut Consumption Sequence
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Evening Peanut Consumption - Evening Snack Sequence | Evening Snack-Evening Peanut Consumption Sequence
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Evening Peanut Consumption-Evening Snack Sequence: First intervention:
  Participants will consume one ounce per day (28 g) of peanuts as an evening snack (i.e., after dinner and before sleep).
  Peanut: Roasted, unsalted peanuts will be purchased from a local grocery store and provided to subjects to consume.
  Second Intervention:
  Participants will consume an isocaloric higher carbohydrate snack as an evening snack (i.e., after dinner and before sleep).
  High carbohydrate snack: Whole wheat crackers will be purchased from a local grocery store and provided to subjects to consume with a spread (e.g. cream cheese or margarine).
- Total: Total of all reporting groups
Arm/Group | Evening Peanut Consumption-Evening Snack Sequence | Evening Snack-Evening Peanut Consumption Sequence | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15) | 43 (15) | 42 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 12 | 14 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Fasting Plasma Glucose
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Evening Peanut Consumption: Evening Peanut Consumption
- Evening Lower-fat Higher-carbohydrate Snack: Evening lower-fat higher-carbohydrate snack
Arm/Group | Evening Peanut Consumption | Evening Lower-fat Higher-carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mg/dL | -0.9 [-2.7 to 0.9] | -0.4 [-2.2 to 1.4]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-fat Higher-carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.7 to 1.6]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.7 to 0.9]
Statistical Analysis 3: Comparison: Evening Lower-fat Higher-carbohydrate Snack; Test type: Other — Change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.2 to 1.4]

2. Secondary Outcome: Fructosamine
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
umol/L | -4.0 [-5.1 to 5.4] | -3.8 [-5.1 to 5.4]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-4.8 to 3.4]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -4, 95% CI 2-sided [-5.1 to 5.4]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-5.1 to 5.4]

3. Secondary Outcome: Fasting Insulin
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
umol/L | -0.2 [-1.5 to 1.0] | -0.8 [-2.1 to 0.5]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-1.2 to 2.1]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.5 to 1.0]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.1 to 0.5]

4. Secondary Outcome: Peripheral Systolic and Diastolic Blood Pressure
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mmHg
  Peripheral systolic within-condition mean difference | 0.4 [-2.5 to 3.3] | -0.3 [-3.1 to 2.6]
  Peripheral diastolic within-condition mean difference | 0.5 [-1.5 to 2.5] | -0.0 [-2.0 to 2.0]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; peripheral systolic BP; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.1 to 4.6]
Statistical Analysis 2: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; peripheral diastolic BP; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.1 to 2.9]
Statistical Analysis 3: Comparison: Evening Peanut Consumption; peripheral systolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.5 to 3.3]
Statistical Analysis 4: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; peripheral systolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.1 to 2.6]
Statistical Analysis 5: Comparison: Evening Peanut Consumption; peripheral diastolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.5]
Statistical Analysis 6: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; peripheral diastolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-2 to 2]

5. Secondary Outcome: Central Systolic and Diastolic Blood Pressure
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mmHg
  Central systolic within-condition mean difference | 0.6 [-1.9 to 3.1] | -0.4 [-2.9 to 2.1]
  Central diastolic within-condition mean difference | 0.5 [-1.5 to 2.6] | -0.4 [-2.4 to 1.6]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; central systolic BP; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.4 to 4.4]
Statistical Analysis 2: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; central diastolic BP; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.7 to 3.3]
Statistical Analysis 3: Comparison: Evening Peanut Consumption; central systolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.9 to 3.1]
Statistical Analysis 4: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; central systolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.9 to 2.1]
Statistical Analysis 5: Comparison: Evening Peanut Consumption; central diastolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.6]
Statistical Analysis 6: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; central diastolic BP change from baseline; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.4 to 1.6]

6. Secondary Outcome: Carotid Femoral Pulse Wave Velocity
Description: Carotid-femoral pulse wave velocity is a measure of arterial stiffness and is determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery.
  Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
m/s | 0.3 [0.1 to 0.6] | 0.1 [-0.1 to 0.3]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.6]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

7. Secondary Outcome: Augmentation Index (%)
Description: A measure of arterial stiffness assessed using a SphymoCor Ecel (Atcor Medical). A higher percentage value is indicative of greater arterial stiffness
  Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: % adjusted to a HR of 75 BPM
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
% adjusted to a HR of 75 BPM | -0.4 [-3.7 to 2.9] | 0.2 [-4.0 to 4.3]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.9 to 3.3]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.7 to 2.9]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.0 to 4.3]

8. Secondary Outcome: LDL Cholesterol
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mg/dL | 2.4 [-2.1 to 6.9] | -2.3 [-6.8 to 2.2]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-1.4 to 9.8]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-2.1 to 6.9]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-6.8 to 2.2]

9. Secondary Outcome: HDL Cholesterol
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mg/dL | 0.6 [-0.6 to 1.8] | 0.6 [-1.6 to 2.3]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.3 to 2.3]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.8]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.6 to 2.3]

10. Secondary Outcome: Total Cholesterol
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mg/dL | 0.1 [-4.9 to 5.1] | -2.7 [-7.8 to 2.3]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-3.8 to 8.2]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-4.9 to 5.1]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-7.8 to 2.3]

11. Secondary Outcome: Triglycerides
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
mg/dL | -17 [-29.1 to -4.8] | -5.7 [-17.1 to 5.7]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-18.3 to 2.8]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -17, 95% CI 2-sided [-29.1 to -4.8]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-17.1 to 5.7]

12. Secondary Outcome: Body Weight
Description: Within-condition mean differences (change from baseline).
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
kg | 0.2 [-0.1 to 1.5] | 0.0 [-0.5 to 0.5]
Statistical Analysis 1: Comparison: Evening Peanut Consumption vs Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 2: Comparison: Evening Peanut Consumption; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 1.5]
Statistical Analysis 3: Comparison: Evening Lower-Fat Higher-Carbohydrate Snack; Test type: Other — change from baseline; Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.5]

13. Secondary Outcome: Microbiota Alpha-diversity
Description: Measured by Faith's Phylogenetic Diversity Score. This is a measure of biodiversity (based on phylogeny). Faith's phylogenetic diversity measures the amount of the phylogenetic tree covered by the bacterial community. It's a sum of the minimum branch lengths. A higher number (more branches), means more richness (more diversity). Increases in Faith's Phylogenetic Diversity is indicative of more richness and diversity but no standard reference range or clinically relevant values have been established.
  Presented as endpoint mean values with IQR
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: Faith's Phylogenetic Diversity Score
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
Number analyzed (Participants) | 50 | 50
Faith's Phylogenetic Diversity Score | 10.4 [7.5 to 13.3] | 10.6 [7.4 to 13.8]

ADVERSE EVENTS:
Time Frame: All 16-wks of trial
Description: No subjects were at risk for serious adverse event or all-cause mortality. Therefore, these were not monitored. Adverse-events (e.g., allergic reactions to study foods) were monitored.
Arm/Group | Evening Peanut Consumption | Evening Lower-Fat Higher-Carbohydrate Snack
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03654651/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03654651/ICF_001.pdf